CLINICAL TRIAL: NCT03257332
Title: The EDFI-Cohort: Determining Early Development of Faecal Incontinence and Anorectal Muscle Function After Curative Surgery for Rectal Cancer.
Brief Title: Determining Early Development of Faecal Incontinence and Anorectal Muscle Function After Surgery for Rectal Cancer.
Acronym: EDFI-Cohort
Status: Withdrawn | Type: Observational
Why Stopped: Not possible to include participants
Sponsor: Slagelse Hospital (Other)
Collaborators: Zealand University Hospital (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Brian Clausen, Physiotherapist and PhD, Slagelse Hospital
Other Study IDs: EDFI-Cohort
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Rectum Cancer; Quality of Life; Faecal Incontinence; Low Anterior Resection Syndrome
Keywords: Rectum cancer; Low Anterior Rectal Syndrome; Anorectal muscle function
MeSH Terms: conditions — Rectal Neoplasms; Encopresis; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EDFI Cohort: Subjects should have received surgery for rectal cancer (low anterior resection).
  Interventions: Procedure: Low Anterior Resection for Rectum Cancer

INTERVENTIONS:
Procedure: Low Anterior Resection for Rectum Cancer — Subjects should have received curative surgery for rectal cancer (low anterior resection) with/with-out adjuvant (radiation/chemo) therapy.
  Other Names: Total mesorectal excision; Partial mesorectal excision

SUMMARY:
Background:

Patients treated for rectal cancer are in high risk of developing poor quality of life and faecal incontinence. Faecal incontinence has a negative impact on quality of life. However, there is limited knowledge on how to prevent it. Known exposures are ; age at surgery, gender, tumor height, pre-operative radiotherapy, surgical technique and temporary stoma. In order to evaluate the underlying mechanisms of faecal incontinence, it is central to evaluate the anorectal muscle function for sensory and motor impairment. Exposures representing different constructs in the biopsychosocial model are likewise likely to be associated with quality of life and faecal incontinence. These exposures include sexual dysfunction, urinary incontinence, fatique, physical inactivity and finding meaning in life. There are to our knowledge, no records on these relationships from prior to surgery to 2 years after. These biopsychosocial exposures are central to include when developing strategies that can prevent poor quality of life and faecal incontinence for patients treated for rectal cancer.

Purpose:

The primary purpose of the EDFI-Cohort study is to determine how several variables (surgical technique, anorectal muscle function, faecal incontinence, urinary incontinence, sexual dysfunction, fatigue, physical activity and finding meaning in life) develop over time and predicts quality of life. Secondary how it predicts LARS-score in patients with rectal cancer from prior to surgery to 2 years after primary treatment.

Methods:

We will include subjects diagnosed with rectal cancer and have received curative surgery (low anterior resection) with/without adjuvant (radiation/chemo) therapy. The cohort aim to recruit all eligible patients in a one year period. We estimate to recruit 70 patients.

Self-reported outcomes will be collected with a series of validated questionnaires that subjects will be asked to complete 6 times during the two year study at 3, 6, 12, 26 78 and 104 weeks. Outcomes include: Quality of life using (EORTC QLQ-C30) (primary outcome), (CR29) and (FA12), bowel related quality of life (LARS-score) (secondary outcome), faecal incontinence (Vaizey score), urinary incontinence (ICIQ-UI), (MLUTS/FLUTS) and (MLUTSsex/FLUTSsex), physical activity level from Danish National Health Profile and finding meaning in life (SOME).

Objective measures will be collected at 6 weeks, 6 months, 12 months and 24 months and include: Anorectal manometry that measures anorectal muscle function and rectal perception, a digital examination of anorectal muscle function using the Digital Rectal Examination Scoring System (DRESS) and the six-minute walk test a measure of submaximal exercise capacity.

We plan to analyze the EDFI-Cohort study as repeated measures with both simple and multiple linear regression models for the continuous data. We plan to adjust for known confounders and variables related to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rectal cancer
* Low anterior resection (e.g. not limited to total mesorectal excision (TME) or partial mesorectal excision (PME))
* Ability to communicate in Danish
* Adults (> 18 years of age)
* American Society of Anaesthesiologists (ASA) score: I-IV.

Exclusion Criteria:

* ASA score of: V-VI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects for the EDFI-Cohort study will be recruited during 2019 and 2020 from Department of Surgery, Slagelse, and Zealand University Hospital, Køge. Subjects need to be diagnosed with rectal cancer and have received curative surgery (low anterior resection) with/without adjuvant (radiation/chemo) therapy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Global health status/quality of life: EORTC QLQ-C30 | 104 weeks
  European Organisation for Research and Treatment of Cancer's generic core set on quality of life (EORTC QLQ-C30)

SECONDARY OUTCOMES:
Low anterior resection syndrome | 104 weeks
  Self-reported questionnaire - Low anterior resection symptom - score (LARS-score)

OTHER OUTCOMES:
Urinary incontinence | 3, 6, 12, 26, 52 and 104 weeks
  International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF)
Urinary incontinence - Urinary symptoms | 3, 6, 12, 26, 52 and 104 weeks
  International Consultation on Incontinence Questionnaire - Male/female Lower Urinary Tract Symptoms (ICIQ-MLUTS og ICIQ-FLUTS)
Urinary incontinence - Sexual dysfunction | 3, 6, 12, 26, 52 and 104 weeks
  International Consultation on Incontinence Questionnaire - Male/female Sexual Matters associated with Lower Urinary Tract Symptoms (ICIQ-MLUTSsex or ICIQ-FLUTSsex)
Global health status/quality of life: EORTC QLQ-C30 | 3, 6, 12, 26 and 52 weeks
  European Organisation for Research and Treatment of Cancer's generic core set on quality of life (EORTC QLQ-C30)
Other subscales than 'global health status/quality of life': EORTC QLQ-C30 | 3, 6, 12, 26, 52 and 104 weeks
  European Organisation for Research and Treatment of Cancer's generic core set on quality of life (EORTC QLQ-C30)
Quality of life - colorectal cancer: EORTC QLQ-CR29 | 3, 6, 12, 26, 52 and 104 weeks
  European Organisation for Research and Treatment of Cancer's colorectal cancer module (EORTC QLQ-CR29)
Quality of life - Fatigue: EORTC QLQ-FA12 | 3, 6, 12, 26, 52 and 104 weeks
  European Organisation for Research and Treatment of Cancer's fatigue module (EORTC QLQ-FA12)
Quality of life - INFO: EORTC QLQ-INFO25 | 3, 6, 12, 26, 52 and 104 weeks
  European Organisation for Research and Treatment of Cancer's information about disease and treatment module (EORTC QLQ-INFO25)
Anorectal muscle function - digital examination | 6, 26, 52 and 104 weeks
  Maximal resting pressure Maximal squeeze pressure Endurance squeeze - max squeeze pressure or longest time Latency (rate of force development), number of rectal muscle contractions/squeezes in 15 sec test.
Anorectal Manometry - pressure | 6, 26, 52 and 104 weeks
  Maximal resting pressure Maximal squeeze pressure Maximal squeeze pressure duration
Anorectal Manometry - capacity | 6, 26, 52 and 104 weeks
  Volume capacity measurements:
  Maximal tolerated volume Conscious rectal sensitivity threshold Conscious rectal sensitivity Constant sensation
Faecal incontinence | 3, 6, 12, 26, 52 and 104 weeks
  Self-reported questionnaire - St. Marks Incontinence score (Vaizey score)
Low anterior resection syndrome | 3, 6, 12, 26 and 52 weeks
  Self-reported questionnaire - Low anterior resection symptom - score (LARS-score)
Physical activity level | 3, 6, 12, 26, 52 and 104 weeks
  physical activity section of the Danish National Health Profile
Finding meaning in life | 3, 6, 12, 26, 52 and 104 weeks
  Sources of Meaning and Meaning in Life Questionnaire (SoMe)
Physical performance | 6, 26, 52 and 104 weeks
  6-Minute Walk test

CONTACTS AND LOCATIONS:
Overall Officials: Søren T Skou, PhD, Study Chair — Slagelse Sygehus; Ismail Gögenur, PhD, Study Chair — Zealand University Hospital
Locations (2):
- Denmark (2):
  - Zealand University Hospital, Køge, Region Sjælland
  - Slagelse Hospital, Slagelse, Region Sjælland

IPD SHARING:
Plan to Share IPD: Undecided
Reseachers whom are interested in study data, are welcome to contact study PI.

REFERENCES:
- [Background] Emmertsen KJ, Laurberg S; Rectal Cancer Function Study Group. Impact of bowel dysfunction on quality of life after sphincter-preserving resection for rectal cancer. Br J Surg. 2013 Sep;100(10):1377-87. doi: 10.1002/bjs.9223. PMID 23939851
- [Background] Lai X, Wong FK, Ching SS. Review of bowel dysfunction of rectal cancer patients during the first five years after sphincter-preserving surgery: a population in need of nursing attention. Eur J Oncol Nurs. 2013 Oct;17(5):681-92. doi: 10.1016/j.ejon.2013.06.001. Epub 2013 Jul 17. PMID 23871359
- [Background] Ma B, Gao P, Song Y, Zhang C, Zhang C, Wang L, Liu H, Wang Z. Transanal total mesorectal excision (taTME) for rectal cancer: a systematic review and meta-analysis of oncological and perioperative outcomes compared with laparoscopic total mesorectal excision. BMC Cancer. 2016 Jul 4;16:380. doi: 10.1186/s12885-016-2428-5. PMID 27377924

DOCUMENTS (2):
  • Study Protocol (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03257332/Prot_000.pdf
  • Informed Consent Form (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03257332/ICF_001.pdf